CLINICAL TRIAL: NCT03815487
Title: Comparison of the Efficacy of Sensor-augmented Pump Therapy Versus Hybrid Closed-loop Glucose Management (MiniMed670G™) in Patients With Type 1 Diabetes at Home in a Randomized Controlled Trial
Brief Title: Comparison of Two Management Systems in Patients With Type 1 Diabetes (Pediatric SmartHome)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PSH-KKB1/ NERP15-028
Record Dates: First submitted 2018-12-05; First posted 2019-01-24 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Patient Care; Drug Therapy
Keywords: pediatrics; type 1 diabetes; insulin pump; closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapy with Hybrid Closed Loop (HCL) (Experimental): The Intervention is the specific function of the Insulin Pump from Medtronic® with the name "MiniMed® 670G (MMT-1780)" to deliver Insulin as medication.
  This Medtronic MiniMed 670G Insulin Pump in Auto Mode is an Hybrid closed loop (HCL) system including an Auto Mode function. It provides as intervention several additional effects concerning automatically insulin delivery by pump: e.g. in case of high values (or predicted) - more insulin will be administered automatically, in case of low values (or predicted) - the insulin infusion will be decreased a suspended and resumed again. The patients will wear the pump continuously.
  Interventions: Device: Medtronic MiniMed 670G Insulin Pump in Auto Mode
- Sensor Augmented Pump (SAP) therapy (Active Comparator): The Intervention is the specific therapy of the Sensor Augmented Insulin Pump "MiniMed® 670G" (MMT-1780) without Auto Mode.
  This Medtronic MiniMed 670G Insulin Pump without Auto Mode' is a Sensor Augmented Pump (SAP) therapy and means the addition of alerts according to high or low glucose values as well as trend arrows showing actual glucose trends to pump therapy. The patients will wear the pump also continuously, but have to respond manually after the alarm. There are no automatically steps from the pump.
  Interventions: Device: Medtronic MiniMed 670G Insulin Pump without Auto Mode

INTERVENTIONS:
Device: Medtronic MiniMed 670G Insulin Pump in Auto Mode — This kind of intervention will be part of the intensified insulin therapy for type 1 diabetic patients. The system will help to keep blood glucose in a defined range by automatic assisted adaption of insulin dosing.the HCL provides a lot more automatic functions to keep glucose in target compared to SAP.
  Other Names: Hybrid Closed Loop (HCL) System
  Arms: Therapy with Hybrid Closed Loop (HCL)
Device: Medtronic MiniMed 670G Insulin Pump without Auto Mode — Sensor augmented pump therapy means the addition of alerts according to high or low glucose values as well as trend arrows showing actual glucose trends to pump therapy. There is no automatic adaption of insulin dosing. The patients must respond manually after alarm or according to the trend arrows.
  Other Names: Sensor Augmented Pump therapy without Auto Mode
  Arms: Sensor Augmented Pump (SAP) therapy

SUMMARY:
Closed loop technology has been shown to reduce both hypoglycemia and hyperglycemia, as well as reduce glycemic variability. Sensor augmented pump (SAP) therapy means the addition of alerts according to high or low glucose values as well as trend arrows showing actual glucose trends to pump therapy. This Hybrid closed loop (HCL) system provides several additional effects compared to SAP therapy: according to actual and predicted sensor glucose values, the insulin therapy can be adopted automatically by pump: in case of high values (or predicted) more insulin will be administered, in case of low values (or predicted) the insulin infusion will be decreased a suspended and resumed again. So the HCL provides a lot more automatic functions to keep glucose in target compared to SAP.

The aim of the current trial is to compare the SAP-therapy with the hybrid closed loop glucose management in patients with type 1 diabetes at home.

DETAILED DESCRIPTION:
Monocentric, randomized, controlled cross-over safety evaluation study. For the study, 20 subjects per age group (small children 2-<9 years, children/adolescents ≥9-14 years) will be enrolled (total n=40). The study is anticipated to last no longer than 6 months from investigational center initiation to completion of all data entry and monitoring procedures. It is estimated that all subjects will be enrolled into the study within approximately 3 months of study start.

* Visit 1 - Day 0: (Subjects come to clinic): Consent, Screening (incl. blood sample) and device training, training to emergency behavior; Pump Start in low glucose suspend mode, alarm settings
* Visit 2 - Week 1: Subjects come to clinic; start Run-in Period and start Sensor Augmented Pump (SAP) therapy without any SmartGuard feature, assessment of AEs; pump will be read out, data stored; subjects will be trained to use the Auto mode, Auto mode will be activated. All subjects will participate in a 11-week study period.
* Visit 3 - Week 2: Subjects are randomized to start with SAP or Hybrid Closed Loop (HCL) therapy and stay with an assigned therapy for next 4 weeks.
* Visit 4 - Week 6: End of Period 1 and start of washout period. Subjects stay in this period with SAP therapy only. Evaluation of past 4 weeks, assessment of AEs
* Visit 5 - Week 7: Period 2 starts. Evaluation of past week, assessment of AEs. SAP group will be using 670G with HCL and HCL group will be using SAP therapy for next 4 weeks.
* Visit 6 - Week 11: End of Study, Subjects come to clinic; evaluation of past 4 weeks, assessment of AEs, HbA1c; pump will be read out, data stored. All study material will be given back.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. At time of screening: Subjects who are 2-14 years are determined by the investigator to be psychologically sound (e.g. no depression, anxiety disorder, traumatic stress disorder) in order to successfully participate in this study
2. Subject has been diagnosed with type 1 diabetes ≥ 1 year Study-specific inclusion criteria

   Subjects will be considered for enrollment in the study if they meet all of the following criteria:
3. Subjects who are 2-14 years are determined by the investigator to have the appropriate, requisite support (family, caregiver or social network) to successfully participate in this study
4. Subject is willing to wear the system continuously throughout the study
5. Subject is willing to perform required sensor calibrations
6. Total daily dose of Insulin >8 U
7. Subject has an A1C value < 12.0% (as processed by Laboratory) at time of screening visit
8. Subject must be on Pump therapy for >3 months prior to Screening
9. Subject may also be on sensor augmented pump therapy.
10. If subject has celiac disease it has been adequately treated as proven by Transglutamase-Antibodies in normal range

Exclusion Criteria:

1. Event of severe hypoglycemia in past 3 months (as per ISPAD Guideline Definition 2014: seizure or loss of consciousness.)
2. Subject is unable to tolerate tape adhesive in the area of sensor placement
3. Subject has any unresolved adverse skin condition in the area of sensor placement (e.g., psoriasis, rash, Staphylococcus infection)
4. Women of child-bearing potential who have a positive pregnancy test at screening or plan to become pregnant during the course of the study
5. Subject has had any of the following new diagnoses within 1 year of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
6. Subject has a clinical significant abnormality (out of reference range, as processed by Laboratory) in thyroid-stimulating hormone (TSH) at time of screening visit
7. Subjects suffering from Morbus Addison, heart failure >NYHA II, chronic pulmonal disease >GOLD II, chronic arterial insuffiency, known cancer disease, diabetic kidney disease, diabetic autonom or peropheral neuropathy
8. Subject tests positive in the drug screen
9. Subject has taken any oral, injectable, or IV steroids within 8 weeks prior time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study; furthermore patients using antipsychotic drugs, antidepressive, ß-blocking agents are not permitted to participate
10. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 4 weeks
11. Subject is currently abusing illicit drugs
12. Subject is currently abusing prescription drugs
13. Subject is currently abusing alcohol
14. Subject is using pramlintide (Symlin) at time of screening
15. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator
16. Subject has elective surgery planned that requires general anesthesia during the course of the study
17. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening
18. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation
19. Subject diagnosed with current eating disorder such as anorexia or bulimia
20. Subject has been diagnosed with chronic kidney disease that results in chronic anemia
21. Subject is on dialysis
22. Subjects known for factitial hypoglycemia or possible suicidal tendencies.
23. Patients who are unwilling or unable to perform a minimum of four blood glucose tests per day.
24. People who are unwilling or unable to maintain contact with their healthcare professional.

Patients whose vision or hearing does not allow cognition of pump signals and alarms.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

PRIMARY OUTCOMES:
Reduction of Sensor Glucose | 6 month
  Time in Range (% of Sensor Glucose 70-180 mg/dL) (SAP period vs Hybrid Closed loop)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Danne, MD, Principal Investigator — Diabetes Centre for Children and Adolescents, Kinderkrankenhaus AUF DER BULT
Locations (1):
- Kinder - und Jugendkrankenhaus AUF DER BULT, Hanover, Germany